CLINICAL TRIAL: NCT06770972
Title: Family Foundations for Individuals Pregnant Via Assisted Reproductive Technology
Brief Title: Family Foundations for Individuals Pregnant Via ART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Eynav Accortt, Associate Professor, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00003470
Record Dates: First submitted 2024-12-17; First posted 2025-01-13 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Assisted Reproductive Technology
Keywords: Assisted Reproductive Technology; mental health outcomes; pregnancy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Foundations immediate enrollment (Experimental): Administer 9 sessions of FF intervention (5 prenatal and 4 postpartum).
  Interventions: Behavioral: Family Foundations
- Family Foundations delayed enrollment (No Intervention): Administer 9 sessions of FF intervention after 3-6 month postpartum. Women will be randomized to either the delayed intervention control or FF.

INTERVENTIONS:
Behavioral: Family Foundations — The FF intervention is 9 sessions, 5 in the prenatal period and 4 in the postpartum period.
  Arms: Family Foundations immediate enrollment

SUMMARY:
The purpose of this study is to help expectant mothers build a coparenting bond and improve communication with a support person (co-caregiver). Participation will include completing two online surveys (one at 12-30 weeks gestation & one at 3 months postpartum), providing two at-home bloodspot collections and returning the collections via mail. Studies suggest that stress increases inflammation. Investigators aim to explore this by collecting a small amount of blood at the first and last session. Participants will also attend 9 virtual one-two hour Family Foundations (FF) intervention sessions (at no cost to participants) with a supportive co-caregiver. Total time commitment will be 18 hours, max, over a 6 month period.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant individuals via ART, at least 18 years of age
2. Have a caregiving partner (e.g. spouse, grandparent; nanny; friend) who will attend sessions
3. Provision of signed and dated informed consent form
4. Stated willingness to comply with all study procedures and availability for the duration of the study
5. English speaking

7. Access to and familiarity with a tablet, smartphone, or computer

Exclusion Criteria:

1. Psychosis
2. Perinatal loss (current) - history of loss is OK
3. Individuals outside of the US
4. Do not have smartphones, tablets, computers (the FF class is virtual)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Depressive Symptoms | From enrollment to the end of intervention at 6 months postpartum
  Change in depression measured by the Edinburgh Postnatal Depression Scale (EPDS). This is a 10-item survey with scores ranging from 0-30 (higher number means more depressive symptoms).
Change in social support | From enrollment to the end of intervention at 6 months postpartum
  Multidimensional Scale of Perceived Social Support (MSPSS): This is a 12-item validated screening tool assessing social support. It has a total score range of 12 to 84, with higher scores indicating higher levels of perceived social support.
Change in Anxiety Symptoms | From enrollment to the end of intervention at 6 months postpartum
  Anxiety symptoms measured by the 5-tiem Overall Anxiety Severity and Impairment Scale (OASIS). The total score on the OASIS ranges from 0 to 20, with higher total indicating more anxiety symptoms.
Change in symptoms of perceived stress | From enrollment to the end of intervention at 6 months postpartum
  Stress measured by the 10-item Perceived Stress Scale (PSS). The PSS score range is 0-40, with higher scores indicating higher levels of perceived stress.
Change in communication | From enrollment to the end of intervention at 6 months postpartum
  Communication Patterns Questionnaire (CPQ): This is a 35 item self-report measure designed to assess the extent to which couples/dyads make use of various interaction strategies during conflict. Each item assesses partners' perception of how likely a certain type of behavior (e.g., both members avoid discussing the problem) occurs when faced with a relationship problem, from 1 (very unlikely) to 9 (very likely). Of the 35 items on the CPQ, 16 are currently used to form four subscales: constructive communication (7 items), self-demand/partner-withdraw (3 items), partner-demand/self-withdraw (3 items), and mutual avoidance (3 items).
Change in symptoms of post-traumatic stress | From enrollment to the end of intervention at 6 months postpartum
  Post-traumatic Stress measured by the 22-item Impact of Event Scale-Revised (IES-R). The IES-R has a score range of 0 to 88, with higher scores indicating more stress.

SECONDARY OUTCOMES:
Change in levels of high sensitivity C-reactive protein (mg/dL) | From enrollment to the end of treatment at 6 months postpartum
  C-reactive protein (CRP) levels are measured with a self-administered blood spot collection kit to indicate inflammation in the body. CRP levels can vary depending on the lab, but here are some general ranges:
  Less than 0.3 mg/dL: Normal for most healthy adults 0.3 to 1.0 mg/dL: Normal or minor elevation 1.0 to 10.0 mg/dL: Moderate elevation More than 10.0 mg/dL: Marked elevation More than 50.0 mg/dL: Severe elevation

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No